CLINICAL TRIAL: NCT04553939
Title: Phase II Study of Neoadjuvant Toripalimab in Combination With Gemcitabine Therapy in Cisplatin Ineligible Stage II-IIIB Bladder Cancer
Brief Title: Neoadjuvant Toripalimab in Combination With Gemcitabine Therapy in Cisplatin Ineligible Local Advanved Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020051314
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: Toripalimab; Neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — toripalimab; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab in Combination With Gemcitabine Therapy (Experimental)
  Interventions: Drug: Toripalimab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 3mg/m2 ivgtt, D1 every 14 days for 2-4 cycles.
Drug: Gemcitabine — Gemcitabine 800mg/m2 ivgtt, D1 every 14 days for 2-4 cycles.

SUMMARY:
This is a pre-surgical study involving subjects with muscle invasive bladder urothelial cancer, who are candidates for cisplatin ineligible neoadjuvant therapy. It is a one-arm phase II study in single center.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* 18-75 years of age on day of signing informed consent.
* Have histologically confirmed muscle invasive disease of the urinary bladder.
* Histology must be urothelial carcinoma (transitional cell carcinoma) or urothelial carcinoma with mixed histology/features.
* Clinical stage II-IIIB and Have a surgical evaluation that documents the plan for multimodality therapy with a consolidative radical cystectomy.
* ECOG 0-1 and good organ function.
* cisplatin ineligible.

Exclusion Criteria:

* A non-surgical approach recommended by the treating urologist due to any reason.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 28 days prior to study registration.
* Has a diagnosis of immunodeficiency or received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Has a known additional malignancy that is progressing or required treatment ≤ 48 months of study registration. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease requiring systemic treatment.
* Has known evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, antibody.
* Has a known history of Human Immunodeficiency Virus.
* Has known active Hepatitis B or Hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
ORR，objective response rate | 3 years
  ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) based upon RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: zhao Shiming, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Balar AV, Castellano D, O'Donnell PH, Grivas P, Vuky J, Powles T, Plimack ER, Hahn NM, de Wit R, Pang L, Savage MJ, Perini RF, Keefe SM, Bajorin D, Bellmunt J. First-line pembrolizumab in cisplatin-ineligible patients with locally advanced and unresectable or metastatic urothelial cancer (KEYNOTE-052): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Nov;18(11):1483-1492. doi: 10.1016/S1470-2045(17)30616-2. Epub 2017 Sep 26. PMID 28967485
- [Background] Wang Z, Till B, Gao Q. Chemotherapeutic agent-mediated elimination of myeloid-derived suppressor cells. Oncoimmunology. 2017 Jun 16;6(7):e1331807. doi: 10.1080/2162402X.2017.1331807. eCollection 2017. PMID 28811975
- [Background] Galluzzi L, Zitvogel L, Kroemer G. Immunological Mechanisms Underneath the Efficacy of Cancer Therapy. Cancer Immunol Res. 2016 Nov;4(11):895-902. doi: 10.1158/2326-6066.CIR-16-0197. PMID 27803050